CLINICAL TRIAL: NCT05200767
Title: The Level of Usual Physical Activity and Its Impact on the Course of COVID-19 in Hospitalized Patients.
Brief Title: Physical Activity and the Course of COVID-19
Status: Completed | Type: Observational
Sponsor: Wroclaw Medical University (Other)
Collaborators: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Edyta Sutkowska, assistant professor, Wroclaw Medical University
Other Study IDs: 1081/2021
Record Dates: First submitted 2022-01-14; First posted 2022-01-21 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: COVID-19; IPAQ; physical activity level; disease severity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Adults aged 18 at the least of any sex and race hospitalized for SARS-CoV-2 infection
  Interventions: Other: completing surveys

INTERVENTIONS:
Other: completing surveys — The level of "usual" physical activity before the disease ( COVID-19- coronavirus disease 2019) will be analysed based on the IPAQ ( International Physical Activity Questionnaire) results.

SUMMARY:
Being active has a beneficial effect on human immunology. Patients hospitalized for COVID-19 (coronavirus disease 2019) will be surveyed for their prior physical activity. In order to show the relationship between the level of usual physical activity and the course of the disease, the following variables will be monitored to express the disease severity: death or transfer to ICU (intensive care unit), or recovery, also the length of hospitalization will be analyzed as a secondary outcome. Depending on the availability of data, the following will also be analyzed: complications other than respiratory failure, C-reactive protein (CRP) and procalcitonin (PCT) levels on admission, and other laboratory parameters, need for oxygen therapy.

DETAILED DESCRIPTION:
The aim of the study is to assess the relationship between the level of physical activity before falling ill with COVID-19 (coronavirus disease 2019) and the severity of the disease. The course of the disease is often surprising and independent of factors that have been selected as poor prognostic factors ( e.g. diabetes, obesity), therefore it is advisable to look for a relationship for those variables that have not yet been analyzed.

Methodology:

To show if the usual physical activity impacts the course of COVID-19 the relationship between the results from the modified, short form of IPAQ (International Physical Activity Questionnaire) and the disease termination (death or transfer to intensive care unit or recovery) as well as the hospitalization length will be analyzed. The modification of the questionnaire is necessary due to the specific course of COVID-19, thus the patients will be asked about the "usual" physical activity before the disease (not about the last 7 days).

After written consent patients (age >= 18) from the temporal hospital, dedicated to COVID-19, will be surveyed with IPAQ. If the patient's condition is too poor, the patient will be able to: provide answers on a different day up to 7 days from discharge from the hospital, or indicate a relative who can answer for him/her. The basic laboratory parameters e.g.: morphology, C-reactive protein, procalcitonin, kidney and liver function, D-dimer, gasometry, and X-rays picture of the lungs will be collected from the patient's medical record if available. Also, information about the type and duration of the used ventilation will be collected if available.

ELIGIBILITY:
Inclusion Criteria:

* age >=18
* confirmed COVID-19 ( coronavirus disease 2019) infection
* hospitalization in the COVID-19 treatment unit

Exclusion Criteria:

* pregnancy;
* inability to complete the questionnaire during hospitalization or up to a week after discharge;
* history of a significant cardiovascular event in the last 6 months (acute coronary syndrome, stroke, amputation, revascularization of peripheral vessels, pulmonary or peripheral embolism of any etiology) if the patient did not complete the rehabilitation process;
* symptomatic chronic respiratory disease not responding to therapy before hospitalization for COVID-19 (or no therapy);
* any dyspnea at rest in the last month before COVID-19;
* injury to the locomotor system in the last month before contracting COVID-19;
* hospitalization in the last month before contracting COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized due to COVID-19 (confirmed COVID-19 infection by PCR method or equivalent diagnostic technique) at the COVID-19 treatment unit
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
death | From the date of admission to hospital until the date of death; assessed up to 5 months
  death due to COVID-19 ( coronavirus disease 2019) complication of the disease
recovery | From the date of admission to hospital until the date of a dismission from the hospital; assessed up to 5 months
  patient discharged home from hospital
transfer to intensive care unit (ICU) | From the date of admission to hospital until the date of transfer to ICU; assessed up to 5 months
  patient moved to intensive care unit

SECONDARY OUTCOMES:
hospitalization length | From the date of admission to hospital until the date of death, transfer to ICU or discharge home;assessed up to 5 months
  days spent in hospital before: death, transfer to ICU or recovery

CONTACTS AND LOCATIONS:
Overall Officials: Edyta Sutkowska, PhD, Study Chair — Wroclaw Medical University
Locations (2):
- Poland (2):
  - Wroclaw Medical University, Wroclaw, Lower Silesian Voivodeship
  - Medical University of Silesia, Bytom, Upper Silesia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication: results of IPAQ, data about the primary and secondary outcomes, laboratory tests, also statistical analysis will be available at the link connected with URN: urn:umed-wroc-prod:UMW9cf7247169fc4d2b8dad0921ad2207fb after publishing; other supporting documents will be available as supplementary materials accompanying the article after publishing
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1. after publication with no time limit for IPD
  2. supplementary materials - depends on the publisher
Access Criteria: 1. under processing of determined- for IPD
  2. according to the publisher law- for the supplementary materials
URL: http://ppm.umed.wroc.pl/info/researchdata/UMW9cf7247169fc4d2b8dad0921ad2207fb/

REFERENCES:
- [Background] Brodin P. Immune determinants of COVID-19 disease presentation and severity. Nat Med. 2021 Jan;27(1):28-33. doi: 10.1038/s41591-020-01202-8. Epub 2021 Jan 13. PMID 33442016
- [Background] Ejaz H, Alsrhani A, Zafar A, Javed H, Junaid K, Abdalla AE, Abosalif KOA, Ahmed Z, Younas S. COVID-19 and comorbidities: Deleterious impact on infected patients. J Infect Public Health. 2020 Dec;13(12):1833-1839. doi: 10.1016/j.jiph.2020.07.014. Epub 2020 Aug 4. PMID 32788073
- [Background] Guo L, Wei D, Zhang X, Wu Y, Li Q, Zhou M, Qu J. Clinical Features Predicting Mortality Risk in Patients With Viral Pneumonia: The MuLBSTA Score. Front Microbiol. 2019 Dec 3;10:2752. doi: 10.3389/fmicb.2019.02752. eCollection 2019. PMID 31849894
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Biernat E, Stupnicki R, Gajewski AK. International Physical Activity Questionnaire (IPAQ) - Polish version. Wych Fiz Sport. 2007;51(1):47-54. (In Polish).

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT05200767/Prot_SAP_ICF_001.pdf